CLINICAL TRIAL: NCT02025933
Title: Title in Norwegian: Ung og Frisk. En Studie av Helseeffekter av Fiskeinntak i Overvektige Barn.
Brief Title: Project Healthy Eating in Children. A Study on the Health Effects of Fish Intake in Overweight Children
Status: Terminated | Type: Observational
Why Stopped: We were unable to recruit a sufficient number of participants
Sponsor: University of Bergen (Other)
Collaborators: The Fisheries and Aquaculture Industry Research Fund (Other)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, Researcher, University of Bergen
Other Study IDs: 2013/541
Record Dates: First submitted 2013-12-17; First posted 2014-01-01 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Children; Age 9-12 years; Overweight (iso-BMI > 25)
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Salmon Group: Participants will eat 75 - 150 grams of salmon for dinner, three times a week for 12 weeks.
  Interventions: Other: Salmon Group
- Cod Group: Participants will eat 75-150 grams of cod for dinner, three times a week for 12 weeks.
  Interventions: Other: Cod Group
- Meat Group: Participants will eat 75-150 grams of mixed meat for dinner, three times a week for 12 weeks.
  Interventions: Other: Meat Group

INTERVENTIONS:
Other: Salmon Group — The children are advised to eat at least 75g of salmon per serving, but no more than 150g
  Groups: Salmon Group
Other: Cod Group — The children are advised to eat at least 75g of cod per serving, but no more than 150g
  Groups: Cod Group
Other: Meat Group — The children are advised to eat at least 75g of meat per serving, but no more than 150g
  Groups: Meat Group

SUMMARY:
It has previously been seen that increased fish intake improves the metabolic health of overweight and obese adults, and animal protein improved metabolic health of obese rats. In this project the investigators will investigate whether increased intake of fish or meat improve metabolic health in children aged 9-12 years as well when replacing processed food. The hypothesis is that increased intake of unprocessed fish or meat will improve metabolic health in children as measured by glucose tolerance, lipid metabolism and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* overweight (iso-BMI > 25)
* 9-12 years
* healthy

Exclusion Criteria:

* diagnosed diseases such as diabetes, CVD, intestinal diseases, arthritis
* prescription medications affecting the metabolism of glucose, lipids or the immune system
* use of supplements containing long chain n-3 fatty acids
* high intake of fish
* food allergy

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cildren aged 9-12 years are invited to participate in the study. The children must be healthy and not use prescription medications that affects lipid metabolism, glucose regulation or the immunesystem.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in metabolic status (glucose, lipids, inflammation) | Baseline and end of intervention period (12 weeks)
  We will investigate any changes in the metabolic status by analyzing parameters affected by changes in glucose homeostasis, lipid metabolism and inflammation.

SECONDARY OUTCOMES:
Body composition | Baseline and end of intervention (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Oddrun A Gudbrandsen, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway